CLINICAL TRIAL: NCT01761175
Title: Comparison of Ultrasound-Guided Single Injection Infraclavicular Block or Ultrasound-Guided Double Injection Axillary Block : A Non-inferiority Randomized Trial
Brief Title: Comparison of Ultrasound-Guided Infraclavicular Block and Ultrasound-Guided Axillary Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Ariane Boivin, MD, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEJ-666
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound-guided infraclavicular block (Active Comparator): Ultrasound-guided single injection infraclavicular block
  Interventions: Procedure: Ultrasound-guided infraclavicular block
- Ultrasound-guided axillary block (Active Comparator): Ultrasound-guided double injection axillary block
  Interventions: Procedure: Ultrasound-guided axillary block

INTERVENTIONS:
Procedure: Ultrasound-guided infraclavicular block — Ultrasound-guided single injection infraclavicular block: using an in-plane technique, 30 mL of mepivacaine 1.5% is injected at the posterior aspect of the artery.
  Arms: Ultrasound-guided infraclavicular block
Procedure: Ultrasound-guided axillary block — Ultrasound-guided double injection axillary block: using an in-plane technique, 25 mL of mepivacaine 1.5% is injected postero-medial to the artery. During needle withdrawal, 5 mL of the same solution is injected close to the musculocutaneous nerve.
  Arms: Ultrasound-guided axillary block

SUMMARY:
The purpose of this study is to compare the rate of complete sensory block at 30 minutes following ultrasound-guided single injection infraclavicular block and ultrasound-guided double injection axillary block. The investigators research hypothesis is that both blocks will show comparable rates of complete sensory block at 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* American Society of Anesthesiologists Class 1 to 3
* Undergoing a surgery at the elbow, forearm, wrist or hand under regional anesthesia

Exclusion Criteria:

* Age less than 18 years
* Body mass index more than 40 kg/m2
* Weight less than 45 kg
* Patient refusal
* Contraindication to regional anesthesia (coagulopathy, local infection at the puncture site, systemic infection)
* Previous neurological deficit in the operated arm
* Severe renal or hepatic failure
* Prior surgery in the axillary or infraclavicular area
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Boivin, MD, Principal Investigator — CHU de Québec; Marie-Josée Nadeau, MD, Principal Investigator — CHU de Québec; Nicolas Dion, MD, Principal Investigator — CHU de Québec; Simon Lévesque, MD, Principal Investigator — CHU de Québec; Pierre C. Nicole, MD, Principal Investigator — CHU de Québec; Alexis F. Turgeon, MD, Msc, Principal Investigator — CHU de Québec
Locations (2):
- Canada (2):
  - Hôpital de l'Enfant-Jésus, Québec
  - Hôpital de Saint-Sacrement, Québec

REFERENCES:
- [Derived] Boivin A, Nadeau MJ, Dion N, Levesque S, Nicole PC, Turgeon AF. Ultrasound-Guided Single-Injection Infraclavicular Block Versus Ultrasound-Guided Double-Injection Axillary Block: A Noninferiority Randomized Controlled Trial. Anesth Analg. 2016 Jan;122(1):273-8. doi: 10.1213/ANE.0000000000001017. PMID 26516803

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound-guided Infraclavicular Block: Ultrasound-guided single injection infraclavicular block
  Ultrasound-guided infraclavicular block: Ultrasound-guided single injection infraclavicular block: using an in-plane technique, 30 mL of mepivacaine 1.5% is injected at the posterior aspect of the artery looking for a crescent-shaped distribution around the artery.
- Ultrasound-guided Axillary Block: Ultrasound-guided double injection axillary block
  Ultrasound-guided axillary block: Ultrasound-guided double injection axillary block: using an in-plane technique, 25 mL of mepivacaine 1.5% is injected in order to obtain a postero-medial spread around the artery. During needle withdrawal, 5 mL of the same solution is injected close to the musculocutaneous nerve.
Period: Overall Study
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Started | 112 | 112
Completed | 112 | 112
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Considering a rate of complete sensory block of 90% for the infraclavicular block and a noninferiority margin of 10%, a sample size of 224 patients was needed to evaluate the noninferiority of the axillary block in comparison to the infraclavicular block at 30 minutes, with a power of 80% and an alpha error of 5% (one-sided hypothesis).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16) | 48 (19) | 50 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 73 | 72 | 145
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (3.8) | 26.4 (4.1) | 25.8 (4.0)
Diabetes [Number; unit: participants] | 9 | 4 | 13
American Society of Anesthesiologists (ASA) preoperative classification [Number; unit: participants] — ASA 1: A normal healthy patient ASA 2: A patient with mild systemic disease with no functional limitation ASA 3: A patient with severe systemic disease and functional limitations
  participants
    ASA 1 | 73 | 60 | 133
    ASA 2 | 37 | 45 | 82
    ASA 3 | 2 | 7 | 9
Site of surgery [Number; unit: participants]
  Hand | 80 | 79 | 159
  Wrist | 23 | 25 | 48
  Forearm | 4 | 2 | 6
  Elbow | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Sensory Block
Description: Complete sensory block is defined by anesthesia to cold sensation in the ulnar, radial, median and musculocutaneous nerves territories.
Time Frame: 30 minutes after block completion
Population: Statistical analyses were conducted according to the intention-to-treat principle
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 112 | 112
percentage of participants | 91 [85 to 95] | 79 [71 to 85]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p < 0.01, Chi-squared

2. Secondary Outcome: Number of Patients With Complete Motor Blocks
Description: Complete motor block is defined by paralysis in the ulnar, radial, median and musculocutaneous nerves territories.
Time Frame: 30 minutes after block completion
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ultrasound-guided Infraclavicular Block: Ultrasound-guided single injection infraclavicular block
  Ultrasound-guided infraclavicular block: Ultrasound-guided single injection infraclavicular block: using an in-plane technique, 30 mL of mepivacaine 1.5% is injected looking for a crescent shape distribution around the artery.
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 112 | 112
percentage of participants | 71 [61 to 79] | 54 [44 to 63]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p < 0.01, Chi-squared

3. Secondary Outcome: Time to Complete Sensory Block.
Description: Complete sensory block is defined by anesthesia to cold sensation in the median, ulnar, radial and musculocutaneous nerves territories.
Time Frame: 5, 10, 15, 20, 25 and 30 minutes after block completion
Population: One patient in the infraclavicular block had an anatomic variation precluding block performance. He was considered a block failure for the primary outcome and for the secondary outcomes of complete motor block and surgical success, on the basis of an intention-to-treat analysis. This patient was not included in the remaining secondary outcomes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 111 | 112
percentage of participants
  5 minutes | 1.8 [0.5 to 7.1] | 4 [1.6 to 9.5]
  10 minutes | 22 [15 to 31] | 21 [14 to 30]
  15 minutes | 51 [43 to 62] | 38 [30 to 49]
  20 minutes | 75 [67 to 83] | 56 [48 to 66]
  25 minutes | 87 [81 to 94] | 70 [62 to 79]
  30 minutes | 91 [84 to 95] | 79 [70 to 85]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p < 0.01, Log Rank

4. Secondary Outcome: Time to Complete Motor Block
Description: Complete motor block is defined by paralysis in the median, ulnar, radial and musculocutaneous nerves territories.
Time Frame: 5, 10, 15, 20, 25 and 30 minutes after block completion
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 111 | 112
percentage of participants
  5 minutes | 0 [0 to 0] | 0 [0 to 0]
  10 minutes | 3.6 [1.4 to 9.4] | 3.3 [1.4 to 7.8]
  15 minutes | 18 [12 to 27] | 14 [9 to 22]
  20 minutes | 41 [32 to 51] | 29 [21 to 38]
  25 minutes | 59 [50 to 68] | 37 [29 to 47]
  30 minutes | 72 [63 to 80] | 53 [45 to 63]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p < 0.01, Log Rank

5. Secondary Outcome: Surgical Block Success Rate
Description: Surgical block success is defined by a nerve block allowing surgery without a rescue block, an infiltration of local anesthetics by the surgeon, administration of analgesics for pain in the surgical field or a general anesthesia.
Time Frame: End of surgery
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 112 | 112
percentage of participants | 93 [86 to 97] | 82 [74 to 89]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p = 0.02, Chi-squared

6. Secondary Outcome: Performance Time of the Nerve Block
Description: Performance time is defined as the sum of imaging time (defined as the time elapsed from the moment the Doppler probe is in contact with the patient to the insertion of the Tuohy needle) and needling time (from the insertion of the needle to its complete removal).
Time Frame: During the performance of the block
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 111 | 112
seconds | 231 [213 to 250] | 358 [332 to 387]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Procedure-related Pain on a Visual Analog Pain Scale
Description: Pain was evaluated by the patient on a visual analog pain scale ranging from 0 (no pain) to 10 (worst pain of their life).
Time Frame: After the nerve block procedure ended, up to 5 minutes.
Population: One patient in the infraclavicular block had an anatomic variation precluding block performance. He was considered a block failure for the primary outcome and for the secondary outcomes of complete motor block and surgical success. This patient was not included in the other secondary outcomes. 3 other participants had missing data for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 109 | 111
units on a scale | 2 [1 to 4] | 2 [1 to 4]
Statistical Analysis 1: Comparison: Ultrasound-guided Infraclavicular Block vs Ultrasound-guided Axillary Block; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Patients With Postoperative Adverse Events Related to Nerve Block
Description: Adverse events were defined by residual numbness, loss of sensitivity or weakness in the operated arm related to block performance or signs of hematoma or infection at the puncture site.
Time Frame: 24 hours after surgery
Population: Four patients in the infraclavicular group and six in the axillary group could not be contacted in the pre-established time frame.
Measure: Number; unit: participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 108 | 106
participants | 0 | 0

9. Secondary Outcome: Number of Patients With Postoperative Adverse Events Related to Nerve Block
Description: as for outcome 8
Time Frame: 1 month after surgery
Population: Eight patients in the infraclavicular group and five in the axillary group could not be contacted in the pre-established time frame.
Measure: Number; unit: participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 104 | 107
participants | 0 | 0

10. Secondary Outcome: Duration of Surgery
Time Frame: The end of surgery
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 111 | 112
minutes | 40 [20 to 55] | 31 [15 to 55]

11. Secondary Outcome: Tourniquet Use
Description: Number of participants who had a tourniquet during the surgery
Time Frame: The end of surgery
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 111 | 112
participants | 84 | 85

12. Secondary Outcome: Duration of Tourniquet
Description: The total time the tourniquet was left inflated
Time Frame: The end of surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Number analyzed (Participants) | 84 | 85
minutes | 37 [27 to 49] | 31 [18 to 50]

ADVERSE EVENTS:
Time Frame: 1 month
Description: Patients were contacted at 24 hours and 1 month following their surgery by an investigator blinded to the technique. Standardized questions were asked about potential complications including signs of injection of hematoma at the puncture site or residual numbness, loss of sensitivity or weakness in the operated limb related to block performance.
Arm/Group | Ultrasound-guided Infraclavicular Block | Ultrasound-guided Axillary Block
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/112
Other Adverse Events (participants affected / at risk) | 3/112 | 1/112
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound-guided Infraclavicular Block (N=112) | Ultrasound-guided Axillary Block (N=112)
Local anesthetic toxicity (Nervous system disorders) | 0 (0) | 1 (1) — Mild signs of local anesthetic toxicity including tinnitus, circumoral numbness, drowsiness, lightheadedness or metallic taste.
Horner syndrome (Nervous system disorders) | 2 (2) | 0 (0) — Ptosis, miosis, and anhidrosis of the side of the face ipsilateral to the block performed
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Hematoma at the puncture site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No